CLINICAL TRIAL: NCT02447705
Title: Replacement of Lamivudine by Telbivudine to Improve Renal Function for Post-transplant Hepatitis B Patients - a Randomized Clinical Trial
Brief Title: Replacement of Lamivudine by Telbivudine to Improve Renal Function
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGMH-IRB-101-3476A3
Record Dates: First submitted 2013-06-03; First posted 2015-05-19 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2013-03

CONDITIONS: Disorder Related to Transplantation; Virus Diseases; Injury Due to Exposure to External Cause
MeSH Terms: conditions — Virus Diseases | interventions — Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamivudine group (No Intervention): continue Lamivudine
- Telbivudine group (Experimental): Telbivudine replaces Lamivudine
  Interventions: Drug: telbivudine

INTERVENTIONS:
Drug: telbivudine — telbivudine replace Lamivudine
  Other Names: sobivo
  Arms: Telbivudine group

SUMMARY:
Nephrotoxicity is one of the adverse effects of lamivudine and dosage of lamivudine has to be reduced if patients' renal function is insufficiency. Telbivudine may improve glomerular filtration rate. This study is to see whether renal function is improved when Lamivudine is replaced by telbivudine in liver transplantation patients.

DETAILED DESCRIPTION:
Liver transplantation is the only effective treatment for the patients with liver failure. Hepatitis B-related liver cirrhosis is the major indication to have liver transplantation in Taiwan. After liver transplantation, prophylaxis of hepatitis B recurrence will be performed by anti-hepatitis B immunoglobulin and anti-viral agents. Currently, lamivudine is the drug the investigators choose to prevent HBV recurrence for many years because it is safe for long-term use. However, nephrotoxicity is one of the adverse effects of lamivudine and dosage of lamivudine has to be reduced if patients' renal function is insufficiency. Recently, the studies on chronic hepatitis B patients showed improvement of glomerular filtration rate for those receiving telbivudine treatment. In this study, the investigators will include our post-transplant HBV patients who have stable liver function, receive lamivudine for prophylaxis of recurrent hepatitis B, and have renal dysfunction in stage II-IV. The patients will be randomized to receive telbivudine or lamivudine continuously at 1:1 ratio. Renal function will be examined at 6 months interval to determine whether renal function is improved. The achievement will determine whether telbivudine is better than lamivudine for the HBV patients with renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Sign inform consent
2. Age is not less than 16 years old.
3. Post liver transplantation patient for HBV-related indication.
4. Chronic hepatitis B transplant patients who are treated by lamivudine for not less than 6 months.
5. eGRF stage 2-4 patients (15<eGFR<90ml)
6. Stable liver function, ALT not more than 2 folds of upper limit.

Exclusion Criteria:

1. Acute rejection with increase CNI dose within a month.
2. Pregnant or nursing.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Renal function measurement | every 2 months, up to 12 months
  Measure eGFR when the patients were enrolled, every 2 months and up to 12 months. The most important time point will be to compare eGRF at 6 month and 12 months after medication conversion to the beginning levels. Renal function is improved if eGRF is better after medication conversion.

SECONDARY OUTCOMES:
hepatitis B recurrence | every 6 months, up to 12 months
  Measure hepatitis B surface antigen every 6 months. If HBs AG appears, hepatitis B recurrence is diagnosed.

REFERENCES:
- [Derived] Lee WC, Wu TH, Wang YC, Cheng CH, Lee CF, Wu TJ, Chou HS, Chan KM, Lee CS. Renal Function Improvement by Telbivudine in Liver Transplant Recipients with Chronic Kidney Disease. Biomed Res Int. 2017;2017:9324310. doi: 10.1155/2017/9324310. Epub 2017 Aug 13. PMID 28884132